CLINICAL TRIAL: NCT02334176
Title: A Prospective, Randomized Comparison Between Single and Double Injection Ultrasound-Guided Axillary Brachial Plexus Block
Brief Title: US Guided Axillary Block With Only One Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Kassab d'Orthopédie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P2014/01
Record Dates: First submitted 2014-12-30; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single injection (Active Comparator): Axillary plexus block performed with single injection dorsally to the artery
  Interventions: Procedure: Ultrasound guided axillary plexus block with 1 injection; Drug: lidocaine 1.5% with epinephrine 5µg/ml
- Double injection (Active Comparator): Axillary plexus block performed with 2 injections: one over musculocutaneous nerve the second one dorsally to the artery
  Interventions: Procedure: Ultrasound guided axillary plexus block with 2 injections; Drug: lidocaine 1.5% with epinephrine 5µg/ml

INTERVENTIONS:
Procedure: Ultrasound guided axillary plexus block with 1 injection — The needle will be advanced until the tip is positioned just dorsal to the artery and 35ml of (lidocaine 1.5% with epinephrine 5µg/ml) is deposited in this location.
  Arms: single injection
Procedure: Ultrasound guided axillary plexus block with 2 injections — The needle will be initially advanced toward musculocutaneous nerve and 7 ml of LA (lidocaine 1.5% with epinephrine 5µg/ml) is deposited around the nerve. The needle will be then advanced until the tip is positioned just dorsal to the artery and 28 ml of (lidocaine 1.5% with epinephrine 5µg/ml) is deposited in this location.
  Arms: Double injection
Drug: lidocaine 1.5% with epinephrine 5µg/ml — 35 ml of lidocaine 1.5% with epinephrine 5µg/ml will be used to perform the axillary plexus block

SUMMARY:
The investigators conducted this prospective, randomized, observer-blinded, non-inferiority trial to compare single perivascular injection to double injection (musculocutaneous nerve and perivascular injection) US guided axillary brachial plexus block.

DETAILED DESCRIPTION:
The investigators have been challenged by the question of whether all a single injection may be enough to successfully perform a axillary plexus block.

Three hundred and twenty patients undergoing elective hand surgery under axillary brachial plexus block will be enrolled into this prospective, randomized, observer-blinded non inferiority trial. Using a computer-generated sequence of random numbers and sealed envelope technique, the patients included will randomly be allocated to receive either single or double injection ultrasound-guided axillary block. The block will be performed with the in-plane technique using a 22 gauge, 50 mm needle and a high frequency linear probe.

In the 2 injection group, the needle will initially be advanced toward musculocutaneous nerve and 7 ml of LA (lidocaine 1.5% with epinephrine 5µg/ml) will be deposited around the nerve. The needle will be then advanced until the tip will be positioned just dorsal to the artery and 28 ml of (lidocaine 1.5% with epinephrine 5µg/ml) will be deposited in this location. In the single injection group using the same LA, and 35 ml will be deposited dorsal the artery.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 year of age, ASA physical status I-III, BMI 25 to 35 Kg/m2

Exclusion Criteria:

* non consents patients, any contraindication to brachial plexus anesthesia (local anesthetic allergy, local infection and coagulopathy), preexisting neuropathy, hepatic or renal failure, pregnancy and surgery in the axillary region.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Success rate | 2 hours after the block performance
  the percentage of patients who successfully complete surgery without any additional anesthesia. Will be assessed at the end of the surgery with an expected average time of 2 hours.
total anesthesia-related time | <30 minutes after the block performance
  The total anesthesia-related time is the sum of performance and onset time (see below).

SECONDARY OUTCOMES:
imaging time | 5 minutes
  The imaging time is defined as the time interval between contact of the US probe with the patient and the acquisition of a satisfactory image of the axillary artery, musculocutaneous nerve and the ulnar nerve. Will be assessed at the end of the imaging process with an an expected average time of 5 minutes.
needling time | 5 minutes
  The needling time is defined as the time interval between the start of the skin weal and the end of LA injection. Will be assessed at the end of local anesthetic injection with an an expected average time of 5 minutes.
number of needle passes | 5 minutes
  The initial needle insertion will count as first pass. Any subsequent needle advancement that will be preceded by a retraction of at least 10mm will count for an extra pass. Thus, the number of needle passes is defined as the sum of the first and the extra needle passes. Will be assessed at the end of local anesthetic injection with an an expected average time of 5 minutes.
Performance time | 10 minutes
  The performance time is defined as the time interval between the first contact of the US probe with the skin and the end of local anesthetic injection. Thus performance time is the sum of the imaging and needling times. Will be assessed at the end of local anesthetic injection with an an expected average time of 10 minutes.
Onset time | every 5 minutes until 30 minutes after the end of the block performance
  The onset time is defined as the time required to obtain a sensorimotor composite score of 14 points (see below).
Sensory blockade | every 5 minutes until 30 minutes after the end of the block performance
  Sensory blockade of the musculocutaneous, median, radial and ulnar nerves will be assessed every 5 minutes until 30 minutes and will be graded according to a 3 point scale using a cold test:0= no block, 1= analgesia (patient can feel touch but not the cold), 2=anesthesia (patient can not feel touch and cold). Sensory blockade of the musculocutaneous, median, radial and ulnar nerves will be assessed on the lateral side of the forearm, the palmar part of the thumb, the lateral part of the dorsum of the hand and the volar side of the fifth finger, respectively.
Motor blockade | every 5 minutes until 30 minutes after the end of the block performance
  Motor blockade will be assessed every 5 minutes until 30 minutes and will be graded on a 3 point scale: 0 = no block; 1 = paresis; 2 = paralysis. Motor blockade of the musculocutaneous, radial, median and ulnar nerves will be evaluated by elbow flexion, wrist extension, thumb opposition, thumb abduction, respectively.
Composite score | every 5 minutes until 30 minutes after the end of the block performance
  The sensorimotor composite score is defined as the sum of the score of each assessed nerve. Overall the maximal sensorimotor composite score will be 16 points. Patient is considered ready for surgery when a minimal composite score of 14 points is achieved, provided the sensory block score was equal or superior to 7 out 8 points.

OTHER OUTCOMES:
paresthesia and numbness | up to 48 hours postoperatively
  Paresthesia and numbness were monitored while performing the block, and up to 48 hours postoperatively.
blood vessel puncture | 10 minutes
  Will be monitored while performing the block, with an expected average time of 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Olfa Kaabachi, M.D, Study Chair — Kassab Institut of orthopedics

REFERENCES:
- [Background] Ay S, Akinci M, Sayin M, Bektas U, Tekdemir I, Elhan A. The axillary sheath and single-injection axillary block. Clin Anat. 2007 Jan;20(1):57-63. doi: 10.1002/ca.20270. PMID 16372345
- [Background] Kjelstrup T, Hol PK, Courivaud F, Smith HJ, Rokkum M, Klaastad O. MRI of axillary brachial plexus blocks: a randomised controlled study. Eur J Anaesthesiol. 2014 Nov;31(11):611-9. doi: 10.1097/EJA.0000000000000122. PMID 25051144
- [Result] Tran DQ, Pham K, Dugani S, Finlayson RJ. A prospective, randomized comparison between double-, triple-, and quadruple-injection ultrasound-guided axillary brachial plexus block. Reg Anesth Pain Med. 2012 May-Jun;37(3):248-53. doi: 10.1097/AAP.0b013e31824611bf. PMID 22354104